CLINICAL TRIAL: NCT01557491
Title: A Randomized Blinded Comparison of Hair Growth Following Either Bevelled or Standard Bi-coronal Scalp Incisions.
Brief Title: Hair Regrowth After Bicoronal Incision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Jeff Fialkov, Craniofacial Surgeon, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 8080808
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Alopecia
Keywords: Alopecia; Coronal Incision; Scar Quality
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Straight Incision (Active Comparator): incision made perpendicular to scalp surface
  Interventions: Procedure: Straight Incision
- Bevelled Incision (Active Comparator): Incision made at 45 degrees to scalp surface
  Interventions: Procedure: Bevelled Incision

INTERVENTIONS:
Procedure: Straight Incision — The incision will be made at a 90 degree angle to the surface of the scalp
  Arms: Straight Incision
Procedure: Bevelled Incision — The Incision will be made at a 45 degree angle to the surface of the scalp.
  Arms: Bevelled Incision

SUMMARY:
Loss of hair growth potential in long surgical scalp incisions can become obvious to the patient and others, given hair's tendency to part along the resulting scar. Bevelling incisions perpendicular to the hair follicle angle may increase hair growth through the scar. However, many factors may be confounders such as wound tension and cauterizing the incision. This study will investigate the effect a bevelled incision has on hair growth preservation compared to a standard incision that incises the skin perpendicular to its surface irrespective of hair follicle angles. Following informed voluntary consent, subjects who require bi-coronal scalp incisions as part of a surgical plan will be enrolled. The right side of this bilateral incision will be randomized to receive either a bevelled or a standard incision and the left side will receive the opposite type. During routine surgical follow-up the hair growth within the scar of the two sides will be recorded for comparison and it is our hypothesis that the side with the bevelled incision will have more hair within the scar.

ELIGIBILITY:
Inclusion Criteria:

* Bicoronal Incision required as part of surgical plan
* Incision within hair-bearing scalp

Exclusion Criteria:

* Previous Bicoronal Incision
* Unfit for Surgery
* Unable to provide informed consent
* Unable to comply with followup
* Preexisting alopecia of scalp
* Cutaneous malignancy of scalp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Hair Regrowth Within the Scar | 12 months
  Hair growth through the scar will be counted at 6 and 12 month followup

SECONDARY OUTCOMES:
Scar Characteristics | 1 year post surgery
  Scars will be rated based on the Vancouver Scar Scale (Sullivan, 1990)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew A Plant, MD, Study Director — University of Toronto Plastic and Reconstructive Surgery
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Camirand A, Doucet J. A comparison between parallel hairline incisions and perpendicular incisions when performing a face lift. Plast Reconstr Surg. 1997 Jan;99(1):10-5. doi: 10.1097/00006534-199701000-00002. PMID 8982181
- [Background] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734